CLINICAL TRIAL: NCT04281667
Title: Mechanical Bowel Preparation and Oral Antibiotics Versus Mechanical Bowel Preparation Only Prior Rectal Surgery - a Prospective, Randomized Controlled Trial
Brief Title: Mechanical Bowel Preparation and Oral Antibiotics Versus Mechanical Bowel Preparation Only Prior Rectal Surgery
Acronym: MOBILE2
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Ville Sallinen, Adj. Prof., Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 14112018
Record Dates: First submitted 2020-02-14; First posted 2020-02-24 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Rectal Adenocarcinoma; Rectum Neoplasm; Rectum Carcinoma; Colorectal Cancer; Colorectal Neoplasms; Colorectal Carcinoma; Surgical Site Infection; Surgery--Complications
MeSH Terms: conditions — Rectal Neoplasms; Colorectal Neoplasms; Surgical Wound Infection | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mechanical Bowel Preparation and Oral Antibiotics (Experimental): Mechanical Bowel Preparation and Oral Antibiotics
  Interventions: Drug: Oral Antibiotics; Drug: Mechanical Bowel Preparation
- Mechanical Bowel Preparation Only (Active Comparator): Mechanical Bowel Preparation Only
  Interventions: Drug: Placebo; Drug: Mechanical Bowel Preparation

INTERVENTIONS:
Drug: Oral Antibiotics — Oral antibiotics (neomycin 1g and metronidazole 1g at 3pm and 11pm the day before surgery)
  Arms: Mechanical Bowel Preparation and Oral Antibiotics
Drug: Placebo — Oral placebos (placebo 1 and placebo 2 at 3pm and 11pm the day before surgery)
  Arms: Mechanical Bowel Preparation Only
Drug: Mechanical Bowel Preparation — Mechanical Bowel Preparation using 2L polyethylene glycol (Moviprep)

SUMMARY:
MOBILE2 is a randomized controlled trial comparing mechanical and oral antibiotic bowel preparation to mechanical bowel preparation only in patients undergoing anterior rectal resection with primary anastomosis. Primary endpoint is Comprehensive Complication Index within 30 days from surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for anterior rectal resection with primary anastomosis

Exclusion Criteria:

* Emergency operation
* Bowel obstruction
* Existing stoma
* Other reason preventing mechanical bowel preparation
* Allergy to neomycin or metronidazole
* Age < 18 years
* Lack of co-operation

Exclusion criteria after randomization:

* Patient did not undergo surgery
* Anterior resection was not performed
* Colonic anastomosis was not performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 604 (Estimated)
Dates: Start 2020-03-18 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2027-10-10 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Complication Index | Within 30 days from surgery
  Comprehensive Complication Index score

SECONDARY OUTCOMES:
Surgical Site Infection | Within 30 days from surgery
  Surgical site infection as defined by CDC
Anastomotic dehiscence | Within 30 days from surgery
  Anastomotic dehiscence
Lenght of hospital stay | Within hospital stay, estimated on average 7 days
  Lenght of hospital stay
Mortality | Within 90 days from surgery
  Mortality
Adjuvant therapy | Within 6 months from surgery
  Patients receiving adjuvant therapy divided by patients needing adjuvant therapy

OTHER OUTCOMES:
5-year overall survival | 5 years from surgery
  5-year overall survival
5-year disease specific survival | 5 years from surgery
  5-year disease specific survival
5-year recurrence free survival | 5 years from surgery
  5-year recurrence free survival
Quality of life (SF-36) | At randomization and at one year from surgery
  Difference in quality of life between baseline and 1 year measured using SF-36
Quality of life (QLQ-C30) | At randomization and at one year from surgery
  Difference in quality of life between baseline and 1 year measured using QLQ-C30
Quality of life (QLQ-CR29) | At randomization and at one year from surgery
  Difference in quality of life between baseline and 1 year measured using QLQ-CR29
Quality of life (LARS) | At randomization and at one year from surgery
  Difference in quality of life between baseline and 1 year measured using LARS
Adverse effects of antibiotics | Within 30 days from surgery
  Adverse effects of antibiotics
Bowel microbiota | Before, at, 6 months, and 1 year after surgery.
  Bowel microbiota

CONTACTS AND LOCATIONS:
Overall Officials: Laura Koskenvuo, MD, PhD, Principal Investigator — Helsinki University Central Hospital; Anna Lepistö, MD, PhD, Study Chair — Helsinki University Central Hospital; Ville Sallinen, MD, PhD, Study Director — Helsinki University Central Hospital
Locations (3):
- Finland (3):
  - Helsinki University Hospital, Helsinki
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: No
Individual deidentified participant data will not be available for sharing. Study protocol will be available.

REFERENCES:
- [Derived] Koskenvuo L, Lunkka P, Varpe P, Hyoty M, Satokari R, Haapamaki C, Lepisto A, Sallinen V. Morbidity After Mechanical Bowel Preparation and Oral Antibiotics Prior to Rectal Resection: The MOBILE2 Randomized Clinical Trial. JAMA Surg. 2024 Jun 1;159(6):606-614. doi: 10.1001/jamasurg.2024.0184. PMID 38506889
- [Derived] Willis MA, Toews I, Soltau SL, Kalff JC, Meerpohl JJ, Vilz TO. Preoperative combined mechanical and oral antibiotic bowel preparation for preventing complications in elective colorectal surgery. Cochrane Database Syst Rev. 2023 Feb 7;2(2):CD014909. doi: 10.1002/14651858.CD014909.pub2. PMID 36748942
- [Derived] Koskenvuo L, Lunkka P, Varpe P, Hyoty M, Satokari R, Haapamaki C, Lepisto A, Sallinen V. Mechanical bowel preparation and oral antibiotics versus mechanical bowel preparation only prior rectal surgery (MOBILE2): a multicentre, double-blinded, randomised controlled trial-study protocol. BMJ Open. 2021 Jul 9;11(7):e051269. doi: 10.1136/bmjopen-2021-051269. PMID 34244284
- [Derived] Koskenvuo L, Sallinen V. Preoperative oral antibiotics in colon surgery. Lancet Gastroenterol Hepatol. 2020 Sep;5(9):801-802. doi: 10.1016/S2468-1253(20)30203-X. No abstract available. PMID 32818460